CLINICAL TRIAL: NCT03547180
Title: Moderators and Mediators of Treatment Change in Panic Disorder and Agoraphobia
Brief Title: Mechanisms of Treatment Change in Panic Disorder and Agoraphobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Collaborators: Boston University (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Heather McClary, Director of Research Compliance, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEUA-2005
Record Dates: First submitted 2016-02-01; First posted 2018-06-06 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Panic Disorder With Agoraphobia
Keywords: Respiration panic; Cognitions; Panic; Treatment; Mediators; Moderators
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Therapy (Active Comparator): The training included four components: (a) educating patients about exacerbating panic symptoms through catastrophic thoughts (vicious cycle), (b) identifying negative cognitions associated with physical sensation triggers of recent panic attacks, (c) practicing replacement of maladaptive cognitions with non catastrophic explanations, and (d) instructing patients in between session exercises during Phase I.
  Interventions: Behavioral: Cognitive Therapy
- Capnometry-Assisted Respiratory Training (Active Comparator): The training included four components: (a) educating patients about the exacerbation of panic symptoms through hypocapnia; (b) directing patients' attention to potentially detrimental respiratory patterns; (c) teaching patients techniques to control their respiration, in particular end-tidal PCO2; and (d) instructing patients in between-session exercises. Between-session exercises using a portable capnometer were to be performed twice a day for 17 min at home or elsewhere during Phase I.
  Interventions: Behavioral: Capnometry-Assisted Respiratory Training
- In-vivo exposure therapy (Other): In this two-phase intervention, patients were randomized (within each site) to first receive five individual, weekly, 1-hr sessions of respiratory skill training (CART) or cognitive skill training (CT; Phase I, Skill Acquisition Training), followed by three weekly sessions of in-vivo exposure (Phase II, Application Training) plus a fourth session at 2-month follow-up.
  Interventions: Behavioral: In-vivo exposure

INTERVENTIONS:
Behavioral: Cognitive Therapy — The training included four components: (a) educating patients about exacerbating panic symptoms through catastrophic thoughts (vicious cycle), (b) identifying negative cognitions associated with physical sensation triggers of recent panic attacks, (c) practicing replacement of maladaptive cognitions with non catastrophic explanations, and (d) instructing patients in between session exercises during Phase I.
  Other Names: CT
  Arms: Cognitive Therapy
Behavioral: Capnometry-Assisted Respiratory Training — The training included four components: (a) educating patients about the exacerbation of panic symptoms through hypocapnia; (b) directing patients' attention to potentially detrimental respiratory patterns; (c) teaching patients techniques to control their respiration, in particular end-tidal PCO2; and (d) instructing patients in between-session exercises. Between-session exercises using a portable capnometer were to be performed twice a day for 17 min at home or elsewhere during Phase I.
  Other Names: CART
  Arms: Capnometry-Assisted Respiratory Training
Behavioral: In-vivo exposure — In this two-phase intervention, patients were randomized (within each site) to first receive five individual, weekly, 1-hr sessions of respiratory skill training (CART) or cognitive skill training (CT; Phase I, Skill Acquisition Training), followed by three weekly sessions of in-vivo exposure (Phase II, Application Training) plus a fourth session at 2-month follow-up.
  Other Names: EXP
  Arms: In-vivo exposure therapy

SUMMARY:
The primary goal of the present study is to identify mechanisms of therapeutic change of two theoretically contrasting therapeutic procedures: The first phase consists of comparing the outcome of the capnometry-assisted breathing therapy (BRT) with cognitive restructuring (CT). During the second phase participants of both interventions will undergo in-vivo exposure.

DETAILED DESCRIPTION:
The primary goal of the present study is to identify mechanisms of therapeutic change of two theoretically contrasting therapeutic procedures: While the rationale of breathing training is based on the assumption that hypocapnea (lower than normal levels of pCO2) is responsible for the development and maintenance of panic disorder, the rationale of cognitive interventions is that the primary mechanism in PD is the cognitive misinterpretation of benign bodily sensations. Further, while breathing training should induce a low-anxiety state (through parasympathetic activation) and, therefore, facilitate habituation to fearful situations, voluntary increases in arousal through hyperventilation (sympathetic activation) has been suggested to facilitate cognitive restructuring during exposure.

In order to study mechanisms that potentially produce clinical improvement, the investigators propose a 2-phase therapeutic intervention: The first phase consists of comparing the outcome of the capnometry-assisted respiratory training (CART) with cognitive restructuring (CT). During the second phase participants of both interventions will undergo in-vivo exposure therapy.

With the data collected from the study, the investigators will test the following hypotheses: (a) CART will produce more reduction in psycho-physiologically relevant measures of panic symptoms compared to CT, while cognitive restructuring will produce more reduction in cognitive parameters of panic symptoms; (b) CART will influence the response to voluntary hyperventilation tests by leading to faster recovery compared to CT. Improvement in respiratory psychophysiology will be correlated with improvement in panic symptom severity; (c) Breathing techniques during exposure will lead to a lower-anxiety state, facilitating but not inhibiting fear extinction as suggested by the safety aid theory

ELIGIBILITY:
Inclusion Criteria:

* A current DSM-IV diagnosis of panic disorder with agoraphobia that is designated by the patient as the most important source of current distress
* Patients must be willing to engage in exposure to fearful situations and sensations

Exclusion Criteria:

* A history of bipolar disorder, psychosis or delusional disorders, current substance abuse or dependence

Medical Exclusion Factors:

* Patients with severe unstable medical illness, or serious medical illness for which hospitalization may be likely within the next three months
* Patients with a history of seizures, angina, myocardial infarction, congestive heart failure, clinically significant arrhythmias, transient ischemic attacks, cerebrovascular accidents, diabetes mellitus, significant asthma, emphysema, or chronic obstructive pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in panic symptom severity assessed by the Panic Disorder Severity Scale/CGI | Pre (Week 0), Mid (Week 5), Post (Week 9), Follow-Up (Week 17)
  Clinician administered; 7 items rated on 0 - 4 scale; scores over 9 suggest the need for formal diagnostic assessment

SECONDARY OUTCOMES:
Cortisol assessments collecting 8 saliva samples per day | Phase II (Weeks 7 - 9)
  was administered to subset of patients for exposure and non exposure days

CONTACTS AND LOCATIONS:
Overall Officials: Alicia E Meuret, Ph.D., Principal Investigator — Southern Methodist University
Locations (1):
- Southern Methodist University, Department of Psychology, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data is available upon request

REFERENCES:
- [Result] Meuret AE, Seidel A, Rosenfield B, Hofmann SG, Rosenfield D. Does fear reactivity during exposure predict panic symptom reduction? J Consult Clin Psychol. 2012 Oct;80(5):773-85. doi: 10.1037/a0028032. Epub 2012 Apr 9. PMID 22486408
- [Result] Meuret AE, Rosenfield D, Seidel A, Bhaskara L, Hofmann SG. Respiratory and cognitive mediators of treatment change in panic disorder: evidence for intervention specificity. J Consult Clin Psychol. 2010 Oct;78(5):691-704. doi: 10.1037/a0019552. PMID 20873904
- [Result] Meuret AE, Hofmann SG, Rosenfield D. Catastrophic Appraisal and Perceived Control as Moderators of Treatment Response in Panic Disorder. Int J Cogn Ther. 2010 Sep 1;3:262-277. doi: 10.1521/ijct.2010.3.3.262. PMID 21088704
- [Result] Meuret AE, Trueba AF, Abelson JL, Liberzon I, Auchus R, Bhaskara L, Ritz T, Rosenfield D. High cortisol awakening response and cortisol levels moderate exposure-based psychotherapy success. Psychoneuroendocrinology. 2015 Jan;51:331-40. doi: 10.1016/j.psyneuen.2014.10.008. Epub 2014 Oct 16. PMID 25462905